CLINICAL TRIAL: NCT01496872
Title: Newborn Cranial Somatic Dysfunction - An Observational Study
Status: Completed | Type: Observational
Sponsor: A.T. Still University of Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 100721-001
Record Dates: First submitted 2011-12-19; First posted 2011-12-21 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Somatic Dysfunction of Cranial Region; Somatic Dysfunction of Cervical Spine; Somatic Dysfunction of Lumbar Spine; Somatic Dysfunction of Sacrum
Keywords: Newborn cranial somatic dysfunction; Newborn observational study; Somatic dysfunction; Cranial strain pattern; Osteopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Two prominent osteopathic physician researchers have studied cranial somatic dysfunction in newborns. Dr Viola Frymann published a paper in 1966 on the presence of somatic dysfunction involving 1250 infants. Dr. Jane Carreiro evaluated 1600 newborns in 1993 for cranial somatic dysfunction. This observational study is intended to continue their work in exploring the presence of cranial somatic dysfunction in newborns. The hypothesis is that there is an increased incidence of somatic dysfunction in newborns birthed by primigravid women and in newborns who experienced a longer second stage of labor.

DETAILED DESCRIPTION:
100 newborns will be assessed for somatic dysfunction of the head, cervical, lumbar, and sacral areas. These findings will be compared to the findings of a standard newborn physical exam and the newborn and maternal history. These records will be reviewed for maternal age, parity, gravity, anesthesia during labor, and estimated gestational age. Birth history and initial newborn assessments will be reviewed for labor augmentation, duration of labor, length of second stage of labor, presence of instrumental delivery(vacuum extraction, forceps delivery, etc.), multiple birth, and presentation at delivery (breech, transverse, or compound presentation). The purpose of the study is to quantify the presence of somatic dysfunction in the newborn. We will assess any relationships between the identified somatic dysfunctions and factors present in the mother's and newborn's medical history.

ELIGIBILITY:
Inclusion Criteria:

* The infant must have been born at NRMC
* The infant must be greater than 6 hours old when enrolled
* The infant must be less than 72 hours old when enrolled
* The mother must volunteer to participate in the study

Exclusion Criteria:

* Born outside NRMC
* Infants who are critically ill will be excluded
* Infants with open spina bifida will be excluded
* Infants with a cleft lip will be excluded
* Infants with a cleft palate will be excluded
* Children who are wards of the state will be excluded

Ages: 6 Hours to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants born at the Northeast Regional Medical Center (NRMC) in Kirksville, MO, between August 1, 2011, and July 31, 2012. The infants must be greater than 6 but less than 72 hours old to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Somatic Dysfunction Scale Score (SDSS) | Newborns were examined between 6 an 72 hours postnatal
  Healthy newborns ages 6 to 72 hours postnatal were physically examined and assessed for somatic dysfunction including asymmetry and motion restriction of the cranium, cervical, lumbar, and sacral regions. Total somatic dysfunction identified was summarized in a somatic dysfunction severity scale (SDSS) by assigning one point for each identified findings. SDSS could range from 0 (no somatic dysfunction) to 34 (all somatic dysfunctions assessed were present). Findings were compared to maternal, newborn, and delivery characteristics. Descriptive analyses and comparisons between the initial newborn assessment and research physical examination were performed.

CONTACTS AND LOCATIONS:
Overall Officials: Erica Waddington, D.O., Principal Investigator — A. T. Still University
Locations (1):
- A. T. Still University/Northeast Regional Medical Center, Kirksville, Missouri, United States

REFERENCES:
- [Background] Frymann V. Relation of disturbances of craniosacral mechanisms to symptomatology of the newborn: study of 1,250 infants. J Am Osteopath Assoc. 1966 Jun;65(10):1059-75. No abstract available. PMID 5178520
- [Background] Carreiro J. Labor, delivery and birth. In: Carreiro, J. An Osteopathic Approach to Children, 2nd ed. Edinburgh: Churchill Livingstone Elsevier, 2009: 131-145.
- [Derived] Waddington EL, Snider KT, Lockwood MD, Pazdernik VK. Incidence of Somatic Dysfunction in Healthy Newborns. J Am Osteopath Assoc. 2015 Nov;115(11):654-65. doi: 10.7556/jaoa.2015.136. PMID 26501758

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2011-07-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT01496872/Prot_SAP_000.pdf
  • Informed Consent Form (2011-07-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT01496872/ICF_001.pdf